CLINICAL TRIAL: NCT04942418
Title: Marginal Adaptation, Shade Matching, and Patient Satisfaction of Polychromatic Feldspathic Laminate Veneer Versus Polychromatic Hybrid Ceramic Laminate Veneer.(Randomize Control Trial)
Brief Title: Marginal Adaptation, Shade Matching, of Polychromatic Feldspathic VS Polychromatic Hybrid Ceramic Laminate Veneer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Kamilia Faisal Abdulkader, (Principal Investigator) PHD candidate in fixed prosthodontic department, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 6221
Record Dates: First submitted 2021-06-22; First posted 2021-06-28 (Actual); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: Adaptation Reaction; Tooth Color; Patient Satisfaction
Keywords: Marginal Adaptation, Shade Matching
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multicolor feldspathic ceramic laminate veneers (Active Comparator): the feldspathic ceramic blocks display the highest translucent properties of all ceramic blocks which make them the first choice in the esthetic zone. esthetic and translucency with polychromatic feature and resilience properties.
  Interventions: Other: Multicolor fieldspathic ceramic laminate veneers.
- Multicolor hybrid ceramic laminate veneers. (Experimental): Multi-shaded blocks have been recently introduced to the market, due to lack of evidence in clinical performance evaluating marginal adaptation and shade matching of the polychromatic newly introduced blocks comparing their different color gradient. Multicolor hybrid ceramic laminate veneers.
  Interventions: Other: Multicolor hybrid ceramic laminate veneers.

INTERVENTIONS:
Other: Multicolor hybrid ceramic laminate veneers. — Multi shaded blocks have been recently introduced to the market, due to lack of evidence in clinical performance evaluating marginal adaptation and shade matching of the polychromatic newly introduced blocks comparing their different color gradient. Multicolor hybrid ceramic laminate veneers.
  Arms: Multicolor hybrid ceramic laminate veneers.
Other: Multicolor fieldspathic ceramic laminate veneers. — the feldspathic ceramic blocks display the highest translucent properties of all ceramic blocks which make them the first choice in the esthetic zone. esthetic and translucency with polychromatic feature and resilience properties.
  Arms: Multicolor feldspathic ceramic laminate veneers

SUMMARY:
The aim of the present study is to evaluate the marginal adaptationو shade matching and patient satisfaction of polychromatic feldspathic porcelain laminate veneer compared to hybrid ceramic multi-color laminate veneer.

DETAILED DESCRIPTION:
PICO P: Population: patients' needs esthetic anterior veneers. I: Intervention: Multicolor hybrid ceramic laminate veneers. C: Comparison: Multicolor feldspathic laminate veneers. O: Outcome: primary: Marginal adaptation. secondary:1 Shade matching 2. Patient satisfaction. S: Study design: Randomized controlled clinical trial. T Time: One year. Research question Will polychromatic hybrid ceramic laminate veneer improve the marginal adaptation, shade matching, and patient satisfaction when compared to polychromatic feldspathic porcelain laminate veneer? Statement of the problem Anterior all-ceramic restoration exhibits esthetic challenge due to color gradient of the tooth nature from cervical to incisor, subsequently, the monochromatic CAD/CAM blocks need external stains which require more time and effort moreover it may leach out over time.

Since the feldspathic ceramic blocks display the highest translucent properties of all ceramic blocks, which make it the first choice in the esthetic zone, on the other hand, it has low strength properties that need careful handling before cementation consequently, the hybrid ceramic overcomes the brittleness characteristic of felspathic ceramics with new material that has comparable esthetic and translucency with polychromatic feature and resilience properties.

Multi-shaded blocks have recently been introducing to the market due to a lack of evidence in clinical performance evaluating marginal adaptation and shade matching of the polychromatic newly introduced blocks comparing their different color gradient. For that, the current study will directly evaluate the shade matching of feldspathic polychromatic porcelain blocks versus hybrid ceramic polychromatic blocks to enhance the multichromatic shade matching of laminate veneers restorations.

Rationale Decision-making for the treatment of esthetic areas performed to achieve highly esthetic outcomes the primary factor for achieving this goal is the material used which, should be of a high shade matching the nature color transition of the natural teeth from cervical to incisal third. Probably the new Enovation of multicolor hybrid ceramic and feldspathic porcelain will solve this problem.

Aim of the study:

The present study aims to evaluate the marginal adaptation, shade matching, and patient satisfaction of polychromatic feldspathic porcelain laminate veneer compared to hybrid ceramic multi-color laminate veneer.

Null hypothesis:

There will be no difference regarding the marginal integrity, shade matching, and patient satisfaction between multicolored feldspathic porcelain anterior laminate veneers and hybrid ceramic multi-color anterior laminate veneers.

III. Methods A) Participants, interventions, and outcomes 9- Study setting: This study will be carried out on patients enrolled from the outpatient clinic in fixed prosthodontics clinic, Faculty of Dentistry, Cairo University 10- Intervention:

10.a.i. Examination and diagnosis:

* Selection and examination of the patients according to inclusion and exclusion criteria proper scaling and polishing procedure will be done
* Primary impressions will take to produce a study cast. The patients will instruct to maintain good oral hygiene by using a toothbrush twice daily.
* Taking a pre-operative professional photo. 10.a.ii. Tooth preparation procedure:

  1. Recording the sulcus depth and gingival condition before preparation.
  2. Conservative tooth preparation will be prepared after local anesthesia has been given as required.
  3. Full coverage preparation will be carried out.

  3. After tooth preparation, adequate 2ry Impression using nonaqueous elastomeric impression materials and bite registration will be taken.

  5. Fabrication of the temporary restoration using composite resin temporary material and cemented using non-Eugenol Zinc Oxide temporary cement.

  10.a.iii. Fabrication and cementation of restoration: Bio-HPP will be supplied in the form of discs to fabricate crown core by CAD/CAM technology then veneered with two veneering techniques; the CAD/ CAM and the manual technique using the viologen system of appropriate shade. The finished Bio HPP crown will cement with adhesive resin cement according to manufacturer instructions.

  10.b. Criteria for discontinuing: Restoration will be removed when there are any signs of leakage, fracture, or severe post-operative pain due to pulpal response and replaced by a temporary restoration cemented with Ca (OH) cement to elevate pain.

  10.c. Strategies to improve adherence to intervention protocol:
* ''In the first visit, a Face to Face adherence session will hold for the patient to be informed about the study steps and how to maintain oral hygiene measures.

Further sessions will occur at the follow-up visits. Participant patients will ask about any problems they are having. Patients will be recalled every three months for one year for follow-up visits.

10.d. Permitted or prohibited interventions: Oral hygiene measures are permitted for enhanced results while using hard toothbrushes or abrasive containing toothpaste after the intervention is prohibited.

11- Outcomes:

- The following assessment surveys (clinical evaluations) will be carried out for both groups: T0 = Preoperative phase: clinical records, periapical radiograph, intraoral photographs, and study casts.

T1 = immediately after final restoration delivery: intraoral photographs. T2 = postoperatively: assessment of the marginal adaptation, shade matching, and patient satisfaction.

ELIGIBILITY:
Inclusion Criteria: All subjects are required to be:

1. patients age range (18-50 years) old, be able to read and sign the informed consent document.
2. Have no active periodontal or pulpal diseases, have teeth with good restorations
3. Psychologically and physically able to withstand conventional dental procedures
4. Patients in a need of anterior veneers.
5. Able to return for follow-up examinations and evaluation

Exclusion Criteria:

1. Patient less than 18 or more than 50 years
2. Patient with active persistent periodontal diseases
3. Patients with poor oral hygiene and uncooperative patients
4. Patients need a smile design for the esthetic zone.
5. Patients in the growth stage with partially erupted teeth
6. Psychiatric problems or unrealistic expectations
7. patient with non-vital teeth.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Estimated)
Dates: Start 2021-12-10 (Estimated); Primary Completion 2024-05-27 (Estimated); Study Completion 2024-11-20 (Estimated)

PRIMARY OUTCOMES:
Marginal adaptation | one year
  Modified USPHS criteria Alfa: Closely adapted (score 1), no visible crevice Bravo: Visible crevice, explorer will penetrate (score 2) Charlie: Crevice in which dentin is exposed (score3) Charlie: Crevice in which dentin is exposed

SECONDARY OUTCOMES:
Shade matching | one year
  Modified USPHS criteria Alfa: Matches tooth (score1) Bravo: Acceptable mismatch (score2) Charlie: Unacceptable mismatch (score3)
Patient satisfaction | one year
  Questionnaire (good and excellent (score1), acceptable (score2), Non-acceptable (score3)

IPD SHARING:
Plan to Share IPD: No